CLINICAL TRIAL: NCT05994716
Title: Effectiveness of Telemedicine in Inflammatory Bowel Disease in Russia
Brief Title: Telemonitoring for IBD Goodness Examination in Russia
Acronym: TIGE-Rus
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department (Other)
Collaborators: Sechenov University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-1
Record Dates: First submitted 2023-07-21; First posted 2023-08-16 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: Inflammatory Bowel Disease; Telemedicine; Telemonitoring
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation group (No Intervention)
- Telemonitoring (Experimental)
  Interventions: Other: Telemonitoring

INTERVENTIONS:
Other: Telemonitoring — A) Monthly completion data on the web platform: 1) SCCAI for Ulcerative colitis and Harvey-Bradshaw index for Crohn disease. 2) IBD disk questionnaire to evaluate disease dynamics. 3) General blood test.
  B) Possibility of online consultation with a gastroenterologist upon request via chat or phone call.
  C) Access to educational information about IBD, necessary lifestyle changes, dietary recommendations;
  D) monthly phone call will be made to each patient from the intervention group to answer any questions or concerns they may have and to interview them according to the checklist.
  Arms: Telemonitoring

SUMMARY:
This is a prospective, randomized study to assess the impact of telemedicine (telemonitoring, tele-education and tele-consultation) on the patients with Inflammatory Bowel Disease (IBD). The main study objective is to evaluate the impact of telemedicine on the quality of life in IBD. The secondary study endpoints are to determine disease activity, the number of IBD relapses, to investigate rate of leukopenia in patients taking azathioprine, to determine medication adherence, psychological well-being and satisfaction with medical care in the telemedicine group in comparison with the face-to-face follow-up group. Moreover, we aim to evaluate association between secondary outcomes and QoL.

It is planned to enroll 64 patients. The study duration is 18 months (12 months - patient enrollment, 6 months - telemonitoring).

The study consists of 3 stages. The first stage is selection of patients with IBD after treatment in the gastroenterology department. The second stage is face-to-face appointment and general recommendations (for the observation group); monthly completion of questionnaires on the web-platform, possibility to contact with doctor via chat or phone call, access to educational information; a monthly phone call to each patient from to answer any questions or concerns they may have and to interview them according to the checklist (for the intervention group). The third stage is the evaluation of IBD activity (re-hospitalization after 6 months), number of IBD relapses, quality of life, frequency of leukopenia in patients receiving azathioprine therapy, medication adherence, psychological well-being and satisfaction with medical care.

DETAILED DESCRIPTION:
Number of volunteers: 64 patients with IBD Study duration: 18 months (12 months - patient enrollment, 6 months - telemonitoring).

Inclusion criteria:

* Age ≥18 years old.
* Signed informed consent.
* Diagnosis: Crohn disease (ICD-10 codes K50.0, K50.1, K50.8, K50.9) and Ulcerative colitis (K51.0, K51.2, 51.3, K51.5, K51.8);
* Treatment in the Gastroenterology Department in Sechenov University Hospital at the moment of trial start.

Exclusion criteria:

* Severe cognitive dysfunction;
* Acute mental illness;
* Lack of technical ability to take part in telemedical intervention (does not have the skills to work with a smartphone, computer, tablet, there is no appropriate technical means);
* Participation in other clinical studies.
* Oncological diseases requiring active treatment.
* Patients who denied signing informed consent.
* Severe decompensation of cogent comorbid ailment;
* Inability to understand written Russian;
* Pregnant individuals.

Outpatient observation with connection to the telemonitoring program - 32 participants.

Outpatient monitoring without connecting to the telemonitoring program - 32 participants.

Study design:

Stage 1: All patients will undergo laboratory tests (including general blood test, C-reactive protein, fecal calprotectin) and instrumental examinations (colonoscopy with biopsy). Computed tomography of the abdomen and pelvis with contrast or magnetic resonance enterography for patients with severe IBD or jejunoileitis will be performed.

After group assignment and signing informed consent, all participants will fill out the following questionnaires:

1. Simple Clinical Colitis Activity Index (SCCAI) questionnaire for patients with ulcerative colitis / Harvey-Bradshaw index (HBI) questionnaire for patients with Crohn disease;
2. World Health Organization's Quality of Life (WHOQOL-26): questionnaire for assessing health-related quality of life;
3. SIBDQ: Short Inflammatory Bowel Disease Questionnaire;
4. Hospital Anxiety and Depression Scale (HADS);
5. Toronto Alexithymia Scale (TAS-26): used to evaluate alexithymia (a risk factor for the development of psychosomatic diseases);
6. Visceral Sensitivity Index (VSI): Special gastroenterological questionnaire to determine the index of visceral sensitivity;
7. PSQ-18: Patient Satisfaction Questionnaire;
8. General Medication Adherence Scale (GMAS) to determine the adherence to the therapy.

Clinical activity of the disease will be measured by Ulcerative Colitis Disease Activity Index (UCDAI) for ulcerative colitis and Crohn's Disease Activity Index (CDAI) for Crohn disease.

All patients will be screened for anxiety, depression, alexithymia and visceral hypersensitivity. A psychiatrist will interview patients with changes in psychological well-being or signs of psychiatric disorders.

Stage 2: Control group patients will receive one face-to-face appointment with gastroenterologist, who will give them recommendations on treatment, surveillance and diet. The standard care for control group will be provided according to the evidence-based guidelines with visits on patient's request.

Telemonitoring group patients will receive authorized access to the personal account on the web platform. The platform contains educational information about IBD, necessary lifestyle changes and dietary recommendations based on international guidelines and education material from Crohn's and Colitis Foundation.

Patients will have to log in to the web platform at least once a month. When the patient logs in to the telemedicine platform they will have to fill out the following data: 1) SCCAI for Ulcerative colitis and Harvey-Bradshaw index for Crohn disease to evaluate clinical activity of the disease during the monitoring; 2) IBD disk questionnaire to evaluate disease dynamics; 3) results of laboratory tests (general blood test, C-reactive protein, fecal calprotectin).

The results of the tests will be available to the health care professionals and the patients. The patients will also have an option of online consultation with a gastroenterologist upon request via chat or phone call. The patients will be instructed to contact a gastroenterologist if they have a recurrence of the disease.

Gastroenterologists will make a phone call to each patient from intervention group with questioning according to the checklist every month. The gastroenterologists will be instructed to provide emergency response in case of critical deviation of health indicators from the limit values or occurrence of complaints indicating the development of an acute condition.

Stage 3: Participants from both groups will be re-hospitalized after 6 months of monitoring. We will evaluate IBD activity according to laboratory and instrumental examinations including general blood tests, C-reactive protein, fecal calprotectin, colonoscopy with biopsy, computed tomography or MR-enterography (for patients with severe IBD or jejunoileitis). Both groups will also have to recomplete all questionnaires to evaluate the study endpoints.

The purpose of this study is to evaluate telemedicine impact in IBD.

ELIGIBILITY:
IInclusion criteria:

* Age ≥18 years old.
* Signed informed consent.
* Diagnosis: Crohn disease (ICD-10 codes K50.0, K50.1, K50.8, K50.9) and Ulcerative colitis (K51.0, K51.2, 51.3, K51.5, K51.8);
* Treatment in the Gastroenterology Department in Sechenov University Hospital at the moment of trial start.

Exclusion criteria:

* Severe cognitive dysfunction;
* Acute mental illness;
* Lack of technical ability to take part in telemedical intervention (does not have the skills to work with a smartphone, computer, tablet, there is no appropriate technical means);
* Participation in other clinical studies.
* Oncological diseases requiring active treatment.
* Patients who denied signing informed consent.
* Severe decompensation of cogent comorbid ailment;
* Inability to understand written Russian;
* Pregnant individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Change the Health-related quality of life in IBD | Upon completion, up to 6 months
  Change the quality of life in IBD according to Short Inflammatory Bowel Disease Questionnaire (SIBDQ). Max score is 70, min score is 10.
  < 50 means poor HRQol; >50 optimal HRQol Higher score means better outcome

SECONDARY OUTCOMES:
Change clinical activity of Crohn Disease (CD) | Upon completion, up to 6 months
  Clinical activity of CD according to Crohn Disease Activity Index (CDAI), which is a 'gold standard' for trials. CDAI consists of questions regarding symptoms, lab tests, extraintestinal complications, general well-being.
  < 150 - remission; 150-300 - mild; 301-450 - moderate; >450 - severe; Lower score means better outcome.
Change clinical activity of Ulcerative Colitis (UC) | Upon completion, up to 6 months
  Clinical activity of UC according to Ulcerative Disease Activity Index (UCDAI) with questions regarding clinical symptoms and endoscopic activity.
  0-2 - remission; 3-6 - mild; 7-10 - moderate; >10 - severe; Lower score means better outcome.
Change General medication adherence | Upon completion, up to 6 months
  Adherence to the prescribed medications, patient compliance, according to General Medication Adherence Scale. 0-26 - non-adherent; 27-33 - adherent.
Change rate of leukopenia in patients taking azathioprine | Upon completion, up to 6 months
  Number of patients taking azathioprine with onset of leukopenia.
Change Satisfaction with medical care | Upon completion, up to 6 months
  Patient satisfaction with healthcare according to Patient Satisfaction Questionnaire - 18 (PSQ-18). Max score is 90, min score is 18.
  Higher score means better outcome.
Change psychological well-being of patients with IBD measured by HADS | Upon completion, up to 6 months
  Change psychological well-being of patients with IBD according to Hospital Anxiety and Depression Scale (HADS). Each item is scored on a response-scale with four alternatives ranging between 0 and 3. Score 8-10 for doubtful cases and ≥11 for definite cases of depression and anxiety.
Change psychological well-being of patients with IBD measured by VSI | Upon completion, up to 6 months
  Change psychological well-being of patients with IBD according to Visceral Sensitivity Index (VSI). Min value is 0, max value is 75. 0-10 - no GI-specific anxiety; 11-30 - moderate GI-specific anxiety; 31 - 75 - severe GI-specific anxiety; Lower score means better outcome.
Change psychological well-being of patients with IBD measured by TAS-26 | Upon completion, up to 6 months
  Change psychological well-being of patients with IBD according to Toronto Alexithymia Scale (TAS-26) questionnaire. 26-62 - no alexithymia; 63-74 - a doubtful case; 75 - 130 - a definitive case. Lower score means outcome.
Change the quality of life in IBD measured by WHOQOL-26 | Upon completion, up to 6 months
  Change the quality of life in IBD according to World Health Organization's Quality of Life (WHOQOL-26) questionnaire. Max score is 100% min score is 0% for each domain.
  Higher score means better outcome.

OTHER OUTCOMES:
To determine Endoscopic activity of UC | Upon completion, up to 6 months
  Endoscopic activity of UC will be measured by Mayo Endoscopic Score (MES). 0 - normal or inactive disease;
  1. - mild disease with erythema, decreased vascular patterns and mild friability;
  2. - moderate disease with marked erythema, absence of vascular patterns, friability and erosions;
  3. - severe disease with spontaneous bleeding and ulceration. Lower score means better outcome.
To determine Endoscopic activity of CD | Upon completion, up to 6 months
  Endoscopic activity of UC will be measured by Simple Endoscopic Score for Crohn's Disease (SES-CD). 0-2 - remission; 3-6 - mild severity; 7-15 - moderate severity; >15 - severe. Lower score means better outcome.
To determine Histological activity of IBD | Upon completion, up to 6 months
  Histological activity of IBD will be measured via binary scale: presence of signs of inflammation in the histological material; no signs of inflammation in the histological material.
General medication adherence differences | Upon completion, up to 6 months
  Change of the adherence to the prescribed medications, interpreted in 5 levels of adherence. 0-10 - poor adherence; 11-16 - low adherence; 17-26 - partial adherence; 27-29 - good adherence; 30-33 - high adherence. Higher score means better outcome.
Change the number of non-scheduled medical encounters | Upon completion, up to 6 months
  Number of unplanned visits to the Physician for IBD symptoms as recorded in electronic health record.
Change the number of surgical interventions | Upon completion, up to 6 months
  Number of surgical interventions for IBD complications as recorded in electronic health record.
Change the number of of hospitalizations | Upon completion, up to 6 months
  Number of unplanned hospital admissions for any reason as recorded in electronic health record.

CONTACTS AND LOCATIONS:
Overall Officials: Yuliya F Shumskaya, Principal Investigator — Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department; Anton V Vladzymyrskyy, PhD, Study Director — Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department
Locations (1):
- Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No